CLINICAL TRIAL: NCT00461162
Title: Dyspnea Self-Management: Internet or Face-to-Face
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCRC 43-09; R01NR008938 (NIH); R01NR008938-01A2 (NIH)
Record Dates: First submitted 2007-04-13; First posted 2007-04-17 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- 1: i-DSMP (Experimental): Internet Dyspnea Self-management Program (i-DSMP)
  Interventions: Behavioral: Internet DSMP
- 2: f-DSMP (Experimental): Face-to-Face Dyspnea Self-management Program (f-DSMP)
  Interventions: Behavioral: Face-to-Face Dyspnea Self-management
- 3: AC (Active Comparator): Attention Control (AC)
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Internet DSMP — Internet Dyspnea Self-management Program (i-DSMP): Education and skills training for dyspnea management; an individualized tailored exercise plan; self-monitoring of exacerbation symptoms and exercise; and reinforcement/personalized feedback for self management. I-DSMP participants will receive their accessing the modules through the website and participating in weekly online group chat sessions with the research nurse and other participants.
  Arms: 1: i-DSMP
Behavioral: Face-to-Face Dyspnea Self-management — Face-to-Face Dyspnea Self-management Program (f-DSMP): Education and skills training for dyspnea management; an individualized tailored exercise plan; self-monitoring of exacerbation symptoms and exercise; and reinforcement/personalized feedback for self management. F-DMSP participants will attend face-to-face group education sessions. The f-DSMP participants will be provide with a hard copy of the education modules and will participate in six 1-hour group sessions for a period of 6 weeks.
  Arms: 2: f-DSMP
Behavioral: Attention Control — 6 Monthly general health education classes and biweekly telephone calls from a health educator.
  Arms: 3: AC

SUMMARY:
Chronic obstructive pulmonary disease, including emphysema and chronic bronchitis, is the fourth most common cause of death and the second leading cause of disability in the United States. COPD is estimated to be responsible for more than 13.4 million physician visits and 13% of hospitalizations nationally. These hospitalizations are usually caused by acute exacerbations characterized by an increase in symptoms including dyspnea or shortness of breath (SOB), cough, wheezing, and sputum production. The significant disability for people with COPD is primarily due to the symptom of dyspnea (shortness of breath) that affects an individual's quality of life more than does the physiological impairment. Despite optimal medical and pharmacological therapy, most people with COPD continue to suffer from chronic and progressive dyspnea and other symptoms of cough and fatigue.

We have previously shown that an individualized face-to-face dyspnea self-management program was effective in improving dyspnea with activities of daily living (ADL), physical functioning, and self-efficacy for managing dyspnea. Using an experimental longitudinal design, the i-DSMP will be compared to the Face-to-Face Dyspnea Self-Management Program (f-DSMP) and to an Attention Control (AC) intervention

DETAILED DESCRIPTION:
At the present time, education about symptom management for patients and treatments, including exercise, are primarily provided within structured and episodic pulmonary rehabilitation (PR) programs. These PR programs are of short duration, are available for only a small percentage of people because they are expensive and not covered by all third party payers, and often require travel by patients who are disabled. Given estimates of 10 to 24 million U.S. adults with COPD,most of who would benefit from PR, only less than 0.1% can be accommodated at any given time. In the US the maintenance or exercise programs following PR are not reimbursed and, therefore, not available for most patients.

A number of self-management programs have been tested in multiple chronic diseases,but there has been less study of self-management programs for patients with COPD. The few self-management programs for COPD that include only education and limited skills training have not significantly improved symptoms. Home-based PR and self-management programs with nurse home visits have been studied and provide a less costly and accessible alternative. Clearly there is a growing need for more accessible and alternative avenues for providing ongoing support and therapy for COPD patients.

The Internet provides a new exciting delivery channel that offers patients with disabilities an opportunity for greater involvement in health care decision-making and unparalleled opportunities to learn, inform, and communicate with one another and for health care providers to support patients' self-management efforts. Several Internet-based studies for other chronic illnesses have increased self-efficacy for symptom management, perception of available support, and patients' involvement in health care decision making, while reducing symptoms and health care costs. The only published study evaluating the use of the internet to support self-management in COPD patients was our pilot study for this proposal. Our study demonstrated an improvement in both self-efficacy and dyspnea with daily activities measures. This study will expand on the findings of our pilot study.

ELIGIBILITY:
Inclusion Criteria:

* Participants will have:

  1. a diagnosis of COPD which is clinically stable (including medications) for at least one month;
  2. spirometry results showing at least mild obstructive disease defined as post bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio <0.70 with FEV1<80% predicted or post-bronchodilator FEV1/FVC ratio <0.60 with FEV1>80% predicted;
  3. ADL limited by dyspnea;
  4. a designated primary care physician;
  5. ability to speak English and sign consent form;
  6. actively using a computer and the Internet;
  7. no formal pulmonary rehabilitation training for at least 12 months;
  8. patients receiving supplemental oxygen will be acceptable if their O2 saturation can be maintained at >80% on <6L/min of nasal oxygen;
  9. understands how to and is able to rate their shortness of breath during exercise;
  10. age > 40 years.

Exclusion Criteria:

* Subjects will be excluded if they have active symptomatic illness (e.g., cancer, left heart failure, ischemic heart disease with known coronary artery or valvular heart disease, psychiatric illness, and neuromuscular disease).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2007-01; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Dyspnea with ADL | 3, 6, and 12 months
Exercise and functional performance | 3, 6, and 12 months
Exercise adherence | 3, 6, and 12 months
Acute COPD exacerbations | 3, 6, and 12 months

SECONDARY OUTCOMES:
Perception of social support | 3, 6, and 12 months
Self-efficacy for exercise and managing dyspnea | 3, 6, and 12 months
Health resource utilization | 3, 6, and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Carrieri-Kohlman, RN, DNSc, Principal Investigator — University of California, San Francisco
Locations (2):
- United States (2):
  - Dyspnea Research Group, Dept. of Physiological Nursing, University of California, San Francisco, San Francisco, California
  - University of Washington, Seattle - Dept. of Biobehavioral Nursing and Health Systems, Seattle, Washington

REFERENCES:
- [Derived] Nguyen HQ, Donesky D, Reinke LF, Wolpin S, Chyall L, Benditt JO, Paul SM, Carrieri-Kohlman V. Internet-based dyspnea self-management support for patients with chronic obstructive pulmonary disease. J Pain Symptom Manage. 2013 Jul;46(1):43-55. doi: 10.1016/j.jpainsymman.2012.06.015. Epub 2012 Oct 13. PMID 23073395